CLINICAL TRIAL: NCT07182240
Title: Pilot Study of Line-Field Confocal Optical Coherence Tomography for Detection of Mohs Micrographic Surgery Margins of Basal Cell Carcinomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I-3839125
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Noninvasive Imaging Procedue -Line-field optical coherence tomography(LC-OCT) (Other): LC-OCT imaging
  Interventions: Device: LC-OCT Imaging

INTERVENTIONS:
Device: LC-OCT Imaging — handheld imaging device will take high resolution images of lesion

SUMMARY:
To assess the feasibility and provide information on the utility of noninvasive line field confocal optical coherence tomography (LC-OCT) for the presurgical assessment of Mohs micrographic surgery sites in patients undergoing removal of cutaneous basal cell carcinomas (BCC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participant must understand the investigational nature of this study and provide written consent prior to receiving any study-related procedure.
* Participant must be clinically eligible for Mohs surgery as determined by their referring dermatologist and the Mohs surgeon.
* The participant must have a BCC with superficial histology or a BCC with multiple histological features that also include superficial histology, which is appropriate for Mohs surgery.

Exclusion Criteria:

* Known or reported allergy to mineral oil, the optical agent used during imaging.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* . Any condition which in the investigator's opinion deems the subject an unsuitable candidate to undergo imaging procedure.
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Number of cases with fully evaluable images | 1.5 years
  cases were the image evaluator can assess the margins based on image quality

SECONDARY OUTCOMES:
Patient interest in study | 1.5 years
  Will be measured by documenting the number of patients offered study participation and the number choosing to participate in the study
Patients overall experience | one office visit - immediately after imaging procedure
  Collect a 3-question questionnaire to document patients experience.
Determine LC-OCT imaging's impact on surgical workflow | To be filled out immediately after finishing Mohs procedure
  Will be assessed by results of imaging assessment questionnaire given to surgeon
Accuracy of LC-OCT findings | 1.5 years
  Will be evaluated by Comparing LC-OCT findings with frozen section histopathological results
Accuracy of LC-OCT in detectng location of tumor | 1.5 years
  will be evaluated by comparing the location of the LC-OCT reported margin positivity to the Mohs map

CONTACTS AND LOCATIONS:
Overall Officials: Gyorgy Paragh, MD, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States